CLINICAL TRIAL: NCT01247038
Title: A Multicentre Prospective Randomised Control Trial to Compare Two Articulating Bearing Surfaces, Ceramic on Metal and Metal on Metal Large Diameter Femoral Heads, as Used in Cementless Primary Hip Arthroplasty
Brief Title: A Multicentre Trial to Compare Two Articulating Bearing Surfaces as Used in Cementless Primary Hip Arthroplasty
Acronym: MagnumCRCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Biomet's focus has changed and we no longer expect further developments
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU33; Biomet UK Healthcare Ltd (Other: Biomet UK Healthcare Ltd)
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Metal-on-Metal Joint Prostheses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metal on ceramic articulation (Experimental): The arm consists of patients with Ceramic femoral heads articulating with metal acetabular cups
  Interventions: Device: Metal on ceramic articulation
- Metal-on-metal (Active Comparator): The arm consists of patients with Metal femoral heads articulating with metal acetabular cups
  Interventions: Device: Metal-on-Metal

INTERVENTIONS:
Device: Metal on ceramic articulation — Metal on ceramic articulation against metal-on-metal articulation using the same Recap Acetabular cup
  Other Names: MagnumC
  Arms: Metal on ceramic articulation
Device: Metal-on-Metal — Metal on Metal articulation
  Other Names: Magnum
  Arms: Metal-on-metal

SUMMARY:
The aim of this study is to demonstrate the non-inferiority of the ceramic-on-metal articulation using large diameter bearings (38mm to 60mm) compared to the metal on metal articulation using the same cup in regards to the composite clinical success (CCS) rate at 2 years postoperatively (delta = 10% minimum clinically significant difference in rates).

DETAILED DESCRIPTION:
This multicentre randomised controlled trial will compare the clinical outcome of the ceramic-on-metal articulation against a metal-on-metal articulation using the same Recap Acetabular cup.

The metal ion release will be evaluated at predetermined postoperative intervals during the first 36 months. A trial will be conducted as a clinical trial in accordance with the Medical Devices Directive 93/42/EEC (2002).

A total of 150 patients have to be recruited from the South African centre (2 groups)

The initial study assessment period will be 48 months; 24 months recruitment and 24 months follow-up. The follow-up reviews will be at 6 weeks, 6 months, 1 year, 2 years and 3 years. A 5 year and 10 year clinical review will also be carried out with all patients.

An assessment of incidences of adverse events and metal ion release concentrations will be made when all patients are at 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip replacement
* Patient with degenerative joint disease (inflammatory or non-inflammatory) or any of the composite diagnoses of osteoarthritis,avascular necrosis, legg perthes, rheumatoid arthritis, diastrophic variant, fracture of the pelvis, fused hip, slipped capital epiphysis, subcapital fractures, traumatic arthritis
* Patients preoperative Harris hip score < 80 points
* Patients with limited co-morbidity - ASA I - III
* Patients with normal urea and electrolyte levels and creatinine levels
* Patients must be able to understand instructions and be willing to return for follow-up
* Patients willing to provide blood and urine samples for metal ion analysis at follow-up

Exclusion Criteria:

* Patient preoperative Harris hip score > 80 points
* Pre-existing metal implants
* Patients with significant co-morbidity - ASSA IV - V
* Dementia and inability to understand and follow instructions
* Neurological conditions affecting movement
* Women younger than 45 years old
* Presence of symptomatic arthritis in other lower limb joints
* Patients requiring smaller than 38mm and larger than 60mm diameter femoral heads
* Patients taking NSAIDs and / all drugs that will affect bone metabolism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07-10 (Actual); Study Completion 2015-07-10 (Actual)

PRIMARY OUTCOMES:
Metal ion concentration in blood and urine | 2 years post operatively
  Metal ion concentration will be determined from patients blood and urine at prescribed intervals

SECONDARY OUTCOMES:
Composite Clinical Score (CCS) rate at 2 years post operative | 2 years post operatively

CONTACTS AND LOCATIONS:
Locations (2):
- Orthopaedic Hospital & Rehabilitation Clinic of "Dr Miroslav Zotovic", Banja Luka, Bosnia and Herzegovina
- Johannesburg Hospital, Parktown, South Africa

IPD SHARING:
Plan to Share IPD: No